CLINICAL TRIAL: NCT01389947
Title: Study of Non Major Microcirculation During Extracorporeal Circulation : Relation Between Endothelial Dysfunction and Digestive
Brief Title: Microcirculation During Extracorporeal Circulation
Acronym: CITRON4
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Loic Barrot, PH, Centre Hospitalier Universitaire de Besancon
Other Study IDs: P/2010/105
Record Dates: First submitted 2011-05-06; First posted 2011-07-08 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Mesenteric Ischemia
Keywords: mesenteric ischemia; extracorporeal circulation; microcirculation; cardiac surgery; IFABP; citrullinemia; glycocalyx; vascular occlusion test; NIRS probe on thenar eminence
MeSH Terms: conditions — Mesenteric Ischemia; Citrullinemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma measurments Tissular oxygen saturation using NIRS probe
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Extracorporeal circulation: Patients who have coronary artery bypass graft performed under extracorporeal circulation
- Heart beating group: Patients who have a coronary artery bypass graft without extracorporeal circulation

SUMMARY:
Digestive tract is supposed to be the motor of multiple organ failure. In ICU patients, mesenteric ischemia appears even when macrocirculatory parameters are controlled especially in our experience in patients coming in ICU after a cardiac surgery. The investigators suppose that microcirculatory failure develops and results in suffering of non major organs like muscle, skin and digestive tracts. In this study the investigators monitor digestive tract with plasmatic IFABP dosage and microcirculatory circulation with NIRS during a VOT and plasma glycocalyx measurements. The population is composed by patients having coronary artery bypass during cardiopulmonary bypass.

The first aim of this study is to show that digestive tract is suffering with the use of extracorporeal circulation and will be assessed with Plasmatic Intestinal Fatty Acid Binding Protein when IFABP will more than 300 pg/ml ; and with citrullinemia when citrullinemia will be less than 20 micromol/L.

The second aim is to investigate link between endothelial dysfunction and digestive tract. Endothelial dysfunction is assessed with tissular oxygen saturation before, during and after a vascular occlusion test of 3 minutes (measurement of basal value, desaturation curve, resaturation curve and hyperemic response by measurement of area under curve). Endothelial glycocalyx and NO pathway will be investigate (see under)

Our objective is to enroll 100 patients. The same study will be done in a group of patients who benefit from coronary artery bypass without extracorporeal circulation to see the effects of extracorporeal circulation support.

DETAILED DESCRIPTION:
Population study is patients who benefit from coronary artery bypass grafting under extracorporeal circulation support during intervention. Extracorporeal circulation result in SIRS. We aim to study digestive tract during this intervention.

There are 5 times of measurements : under stable hemodynamic conditions and after beginning of anesthesia, just at the end of extracorporeal circulation, about 15 minutes following aortic unclamping and at the end of the Protamine perfusion, about 90 minutes after the end of extracorporeal circulation and the last time measurement 24 hours later.

At each time measurement are done : blood samples to measure Intestinal Fatty Acid Binding Protein, Citrullinemia that are markers for digestive suffering ; blood samples for measurement of Syndecan 1 CD 138 and Heparan Sulfate, two markers of shedding of the endothelial glycocalyx; blood samples for measurement of NOx and GMPc to assess the NO pathway ; measurement of tissular oxygen saturation with a NIRS probe, before, during and after a vascular occlusion test of 3 minutes. Blood samples for hemoglobin, platelets, coagulation evaluation, urea, creatininemia, liver enzymes and pancreatic enzymes will be done at each time.

The vascular occlusion test is done the day before the surgery when patient is awake without any exercise. This is a reference measurement.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery bypass grafting without any other surgery
* surgery made under extracorporeal circulation
* the same surgeon is operating each time

For the heart beating group, inclusion criteria are :

* coronary artery bypass grafting without any other surgery
* surgery performed under "heart beating" conditions.
* no matter about the surgeon that perform surgery

Exclusion Criteria:

* age under 18
* pregnancy
* refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need surgical revascularization of coronary arteries. Patients can not not benefit of percutaneous coronary intervention and need a cardiac surgery of coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proving that digestive failure appears with extracorporeal circulation for cardiac surgery and is more frequent than the 1 to 3 % percent admitted in precedent studies using clinical endpoints. | 24 hours
  Digestive suffering will be assessed by clinical measurment (pain, vomiting), classical biologic measurment and new specific measurment (intestinal fatty acid binding protein : IFABP and citrullinemia. Plasmatic IFABP of more than 300 pg/ml and citrullinemia of more than 20 micromol/L are used as cut-off to define intestinal failure.
  Microcirculatory will be assessed via a Near InfraRed Spectroscopy (NIRS) probe ajusted on the thenar eminence for the tissular oxygen saturation measurment before, during and after a vascular occlusion test of 3 minutes.

SECONDARY OUTCOMES:
Study links between endothelial impairment and digestive suffering | 24 hours
  Digestive suffering was define before.
  Endothelial impairment is define using :
  * Tissular Oxygen Saturation during vascular occlusion test. The reasturation curve represents endothelial vasodilatory capacities
  * Elevation of Syndecan and Heparan shows the shedding of endothelial glycocalyx We will study the links and the correlation between syndecan and heparan elevation with diminution of resaturation curve and digestive suffering NOx and GMPc will help us for the interpretation of NIRS curves.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Manzon, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Jean Minjoz, Besançon, Franche-Comté, France